CLINICAL TRIAL: NCT03668223
Title: The Promoting Resilience in Stress Management (PRISM) Intervention: a Multi-site Randomized Controlled Trial for Adolescents and Young Adults With Advanced Cancer
Brief Title: The PRISM Intervention: a Multi-site Randomized Controlled Trial for Adolescents and Young Adults With Advanced Cancer
Acronym: PRISM-AC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dana-Farber Cancer Institute (Other)
Collaborators: Children's Hospital Los Angeles (Other); Baylor College of Medicine (Other); University of Pittsburgh Medical Center (Other); Seattle Children's Hospital (Other); National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Abby Rosenberg, Principal Investigator, Dana-Farber Cancer Institute
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: 22-653; STUDY00001229 (Other: Seattle Children's Hospital); R01CA222486 (NIH)
Record Dates: First submitted 2018-08-15; First posted 2018-09-12 (Actual); Results first posted 2024-10-24 (Actual); Last update posted 2025-12-05 (Actual); Status verified 2025-12

CONDITIONS: Cancer; Quality of Life; Anxiety; Depression; Hope; Coping Skills; Communication
MeSH Terms: conditions — Neoplasms; Anxiety Disorders; Depression; Communication

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Promoting Resilience in Stress Management (PRISM) (Experimental): Resilience Skills Training
  Interventions: Behavioral: Promoting Resilience in Stress Management (PRISM)
- Usual Care (No Intervention): Standard psychosocial care

INTERVENTIONS:
Behavioral: Promoting Resilience in Stress Management (PRISM) — Manualized skills training targeting resilience resources: stress-management, goal-setting, cognitive reframing, and meaning-making
  Arms: Promoting Resilience in Stress Management (PRISM)

SUMMARY:
Multi-Site Randomized Controlled Trial testing the efficacy of the Promoting Resilience in Stress Management (PRISM) intervention among Adolescents and Young Adults with Advanced Cancer

DETAILED DESCRIPTION:
Among patients with cancer and their families, early integration of palliative care may improve quality of life. This is particularly important for Adolescents and Young Adults (AYAs) because their distinct developmental challenges related to identity, relationships, and vocation may add to the burden of cancer. Among AYAs with advanced cancer, most understand that they may die and report that discussing end-of-life preferences, goals, and fears would be helpful; however, only 53% engage in such conversations. While national guidelines call for integrated palliative care in AYA oncology, developmentally targeted, evidence-based interventions designed to meet psychosocial and communication needs are lacking.

A potential barrier to improving the experiences of AYAs with advanced cancer may be their limited opportunities to develop "resilience resources" such as stress-management, goal-setting, positive reframing, and meaning-making skills. These resources may mitigate negative outcomes, facilitate engagement in goals of care discussions, and improve quality of life. Furthermore, promoting these resources among AYAs may give them the tools to more successfully navigate the challenges of the cancer experience.

Our research program is built on the central hypothesis that promoting resilience resources will improve psychosocial well-being. Over a series of studies, we developed a conceptual framework of resilience in pediatric cancer, affirmed associations between resilience resources and outcomes, and developed a novel resilience resources intervention (Promoting Resilience in Stress Management, PRISM). PRISM is a manualized, skills-based training program comprised of four 30-60 minute, in-person, one-on-one sessions plus a facilitated parent/caregiver/spouse/significant other family-meeting.

We completed a pilot Randomized Controlled Trial (RCT) to test the efficacy of PRISM among 100 AYAs, 6-months following their diagnosis of new (n=73) or recurrent (n=27) cancer. Results suggest PRISM is feasible, highly acceptable, and associated with increased patient-reported resilience as well as key clinically significant patient-centered outcomes such as quality of life and psychological distress. Subgroup analyses comparing patients with advanced cancer to those with new cancer suggested differentially stronger positive effects in the advanced cancer group, raising a hypothesis to be tested in dedicated trials. However, qualitative feedback from patients with advanced cancer suggested refinements targeting hopes, worries, and contextual meaning-making might strengthen PRISM's usefulness.

The overall objective of this project is to refine PRISM to meet the distinct needs of AYAs with Advanced Cancer. We will first adapt and iteratively test the existing PRISM based on established guidelines for intervention development. Then, we will conduct a multi-site randomized controlled trial to test the efficacy of a new PRISM for Advanced Cancer (PRISM-AC). Findings will inform the development of larger dissemination studies and standards of AYA end-of-life and palliative care. Ultimately, this research has the potential to reduce the burden of cancer in a highly vulnerable population.

ELIGIBILITY:
Inclusion Criteria:

* Age 12-24 years
* Diagnosed with advanced cancer: progressive, recurrent, refractory disease or any diagnosis with estimated overall survival <50% at least 2 weeks prior to enrollment
* Able to speak English
* Able to read English or Spanish
* Cognitively able to participate in interviews

Exclusion Criteria:

* Patient Refusal
* Parent Refusal (if patient <18 years-old)

Ages: 12 Years to 24 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 195 (Actual)
Dates: Start 2019-04-15 (Actual); Primary Completion 2024-01-23 (Actual); Study Completion 2025-10-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Abby R Rosenberg, MD, MS, MA, Principal Investigator — Dana-Farber Cancer Institute
Locations (5):
- United States (5):
  - Children's Hospital Los Angeles, Los Angeles, California
  - Dana Farber Cancer Institute, Boston, Massachusetts
  - University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania
  - Texas Children's Hospital, Houston, Texas
  - Seattle Children's Hospital, Seattle, Washington

IPD SHARING:
Plan to Share IPD: Yes
The Dana-Farber / Harvard Cancer Center encourages and supports the responsible and ethical sharing of data from clinical trials. De-identified participant data from the final research dataset used in the published manuscript may only be shared under the terms of a Data Use Agreement. Requests may be directed to Sponsor Investigator or designee. The protocol and statistical analysis plan will be made available on Clinicaltrials.gov only as required by federal regulation or as a condition of awards and agreements supporting the research.
Supporting Information: Study Protocol, SAP
Time Frame: Data can be shared no earlier than 1 year following the date of publication
Access Criteria: DFCI - Contact the Belfer Office for Dana-Farber Innovations (BODFI) at innovation@dfci.harvard.edu

REFERENCES:
- [Derived] Rosenbaum ARP, Ream M, Fladeboe KM, Lau N, Yi-Frazier JP, Rosenberg AR. Examining Sociodemographic Differences in Response to Resilience Coaching for Adolescents and Young Adults Receiving Hematopoietic Cell Transplantation-A Post Hoc Analysis of the PRISM Intervention. Pediatr Blood Cancer. 2025 Nov;72(11):e31998. doi: 10.1002/pbc.31998. Epub 2025 Aug 31. PMID 40887863
- [Derived] O'Daffer A, Comiskey L, Scott SR, Zhou C, Bradford MC, Yi-Frazier JP, Rosenberg AR. Protocol for the promoting resilience in stress management (PRISM) intervention: a multi-site randomized controlled trial for adolescents and young adults with advanced cancer. BMC Palliat Care. 2023 May 16;22(1):60. doi: 10.1186/s12904-023-01179-4. PMID 37189149
- [Derived] O'Daffer A, Comiskey L, Scott SR, Zhou C, Bradford MC, Yi-Frazier JP, Rosenberg AR. Protocol for The Promoting Resilience in Stress Management (PRISM) Intervention: a multi-site randomized controlled trial for adolescents and young adults with advanced cancer. Res Sq [Preprint]. 2023 Apr 7:rs.3.rs-2748874. doi: 10.21203/rs.3.rs-2748874/v1. PMID 37066150

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Promoting Resilience in Stress Management (PRISM) | Usual Care
Started | 99 | 96
Completed | 69 | 76
Not Completed | 30 | 20
Not completed — Death | 10 | 5
Not completed — Lost to Follow-up | 12 | 12
Not completed — Withdrawal by Subject | 8 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Promoting Resilience in Stress Management (PRISM) | Usual Care | Total
Number analyzed (Participants) | 99 | 96 | 195
Age, Continuous [Mean (Standard Deviation); unit: years] | 16.51 (3.79) | 16.51 (3.99) | 16.51 (3.88)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 43 | 52 | 95
  Male | 56 | 44 | 100
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 40 | 37 | 77
  Not Hispanic or Latino | 55 | 59 | 114
  Unknown or Not Reported | 4 | 0 | 4
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 1 | 2
  Asian | 5 | 5 | 10
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 9 | 7 | 16
  White | 58 | 62 | 120
  More than one race | 22 | 19 | 41
  Unknown or Not Reported | 4 | 2 | 6
Region of Enrollment [Number; unit: participants]
  United States | 99 | 96 | 195
Pediatric Quality of Life Cancer Module [Mean (Standard Deviation); unit: units on a scale] — Pediatric Quality of Life (PedsQL) Cancer Module - This scale was designed to assess pediatric cancer-specific health related quality of life. This is a 27 item scale, with each item rated on a 5-point Likert scale where 0=never and 4=almost always. Higher scores represent better health-related quality of life. Scale range is 0-100.
  units on a scale | 65.12 (15.78) | 63.53 (16.16) | 64.34 (15.95)
Connor-Davidson Resilience Scale [Mean (Standard Deviation); unit: units on a scale] — The Connor-Davidson Resilience scale is used to assess inherent resilience. This is a 10-item instrument with higher scores indicating higher resilience. Each item consists of a 5-point Likert scale for a total of 40 points. The scale range is 0-40.
  units on a scale | 27.34 (7.41) | 29.05 (8.45) | 28.18 (7.96)

OUTCOME MEASURES:

1. Primary Outcome: Pediatric Quality of Life Cancer Module
Description: Pediatric Quality of Life (PedsQL) Cancer Module -This scale was designed to assess pediatric cancer-specific health related quality of life. This is a 27 item scale, with each item rated on a 5-point Likert scale where 0=never and 4=almost always. Higher scores represent better health-related quality of life. Scale range is 0-100.
Time Frame: 3-months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Promoting Resilience in Stress Management (PRISM) | Usual Care
Number analyzed (Participants) | 69 | 76
score on a scale | 66.89 (18.07) | 68.41 (18.07)

2. Secondary Outcome: Hospital Anxiety and Depression Scale (HADS) Total Score
Description: The Hospital Anxiety and Depression Scale total score is a 14 items scale on a 4-point Likert scale (range 0-3). It is designed to measure anxiety and depression. The total score is the sum of all 14 items, ranging from 0-42. Higher scores indicate higher total anxiety/depression.
Time Frame: 3-months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Promoting Resilience in Stress Management (PRISM) | Usual Care
Number analyzed (Participants) | 69 | 76
score on a scale | 8.27 (6.79) | 9.94 (7.77)

3. Secondary Outcome: Snyder Hope Scale
Description: Hope: The Snyder "Hope" Scale measures "the overall perception that one's goals can be met." The instrument scored on an 8-point Likert scale (score range 0-64). Higher scores imply greater levels of hopeful thought patterns.
Time Frame: 3-months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Promoting Resilience in Stress Management (PRISM) | Usual Care
Number analyzed (Participants) | 69 | 76
score on a scale | 48.06 (12.15) | 46.89 (14.46)

4. Secondary Outcome: Connor Davidson Resilience Scale
Description: Resilience: The Connor-Davidson Resilience Scale (CD-RISC) measures inherent resiliency. This is a 10-item scale ranging from 0-40 where higher scores reflect greater perceived resilience.
Time Frame: 3-months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Promoting Resilience in Stress Management (PRISM) | Usual Care
Number analyzed (Participants) | 69 | 76
score on a scale | 28.05 (7.94) | 27.45 (10.16)

ADVERSE EVENTS:
Time Frame: 1 year
Description: All-cause mortality was tracked. Other serious adverse events that were reported included the observation of significant or unexpected distress (via distressed behaviors or verbalizations as noticed by the interventionist) during the delivery of the intervention, and was defined by needing additional reporting or follow-up.
Arm/Group | Promoting Resilience in Stress Management (PRISM) | Usual Care
All-Cause Mortality (participants affected / at risk) | 10/99 | 5/96
Serious Adverse Events (participants affected / at risk) | 0/99 | 0/96
Other Adverse Events (participants affected / at risk) | 0/99 | 0/96

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-04-17): https://cdn.clinicaltrials.gov/large-docs/23/NCT03668223/Prot_SAP_000.pdf